CLINICAL TRIAL: NCT03996564
Title: Battlefield Acupuncture for Acute/Subacute Back Pain in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kyle Johnston, Principal Investigator, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2016.017d
Record Dates: First submitted 2018-09-07; First posted 2019-06-25 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Low Back Pain, Mechanical
Keywords: Battlefield Acupuncture; Auricular Acupuncture; Complementary Alternative Medicine; Military, Service Members; Emergency Medicine; Back Pain; Acute Back Pain; Chronic Back Pain; Alternative Medicine,
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Acetaminophen; Diclofenac; Diazepam; Hydrocodone; oxycodone-acetaminophen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Active Comparator): Battlefield Acupuncture (BFA) has a structured administration sequence that was utilized to limit any variability between investigators administering the treatment. The BFA technique has been suggested that the needles are placed not just in an acupoint but actually "acupoint zones." BFA utilizes one to ten (maximum five points per ear) ASP semi-permanent gold needles® placed in one or both ears. The ASP Gold needle® is a sterile device which inserts a small 2 mm needle into the auricle. It is comprised in single-needle applicator ensuring ease of insertion combined with excellent precision. The needles remain in the ear and fall out spontaneously as early as two hours and up to seven days. After administration of the BFA, if subjects felt that their pain was not controlled based on verbal response, rescue medication could be administered to control pain to a tolerable level for discharge.
  Interventions: Device: Battlefield Acupuncture
- Standard Care Group (Active Comparator): Participants randomized to the standard care group were treated with one, or a combination of selected medications to include oral Acetaminophen 500mg-1000mg, Diclofenac 50mg-75 mg orally, Diazepam 5mg-10 mg intravenous or oral, Hydrocodone 5mg/325mg-10mg/650mg mg oral, or intramuscular Ketorolac 30mg-60 mg, as deemed appropriate by the treating investigator (medical provider). Standard treatment was administered by the investigators based on the patient's presentation and driving status as many of the medications cannot be administered if the subject would operate a vehicle. No standardized algorithm was specified and the route and dose of medications was administered at the provider's discretion. After administration of the traditional standard care medications, if subjects felt their pain was not controlled based on verbal responses, rescue medication would be given to control pain to a more tolerable level for discharge.
  Interventions: Drug: Acetaminophen; Drug: Diclofenac; Drug: Diazepam; Drug: Hydrocodone; Drug: Ketorolac

INTERVENTIONS:
Device: Battlefield Acupuncture — 1-10 needles inserted in systematic nature as described by Battlefield acupuncture protocol.
  Arms: Acupuncture Group
Drug: Acetaminophen — Acetaminophen 500mg-1000mg,
  Other Names: Tylenol
  Arms: Standard Care Group
Drug: Diclofenac — Diclofenac 50mg-75 mg orally
  Other Names: Voltaren
  Arms: Standard Care Group
Drug: Diazepam — Diazepam 5mg-10 mg intravenous or oral
  Other Names: Valium
  Arms: Standard Care Group
Drug: Hydrocodone — Hydrocodone 5mg/325mg-10mg/650mg mg
  Other Names: Norco
  Arms: Standard Care Group
Drug: Ketorolac — oral, or intramuscular Ketorolac 30mg-60 mg
  Other Names: Toradol
  Arms: Standard Care Group

SUMMARY:
The randomized controlled study aims was to investigate the pain control of Battle Field Acupuncture as Primary or Adjunctive Treatment in Back Pain (Acute Musculoskeletal pain) in the (acute pain setting) Emergency Department vs stand of care pain medications.

DETAILED DESCRIPTION:
Purpose: To evaluate the effectiveness of Battlefield Acupuncture versus standard care (medicinal therapy) in an Emergency Room setting for acute/subacute back pain using the Visual Analog Scale (VAS) and Numeric Rating Scale (NRS) to determine changes in pain levels. Secondary outcomes will include performance using the back pain functional scale (BPFS), satisfaction of treatment, and the need for further pain medication after discharge from the emergency department.

Design and Methods: A prospective, randomized control trial, (un-blinded, non-placebo controlled) with convenience sampling based on scheduled clinical shifts in the Emergency Department.

The population consisted of active duty service members and Department of Defense beneficiaries (dependents and retirees) at the DoD's sole Level I trauma center, San Antonio Military Medical Center Emergency Department with acute/subacute, or acute/subacute on chronic back pain as the chief complaint. The participants studied age range was from 18-55 years old without concern for pathological back pain.

Subjects were selected based on their chief complaint identified by the triage nurse. A randomized convenience sampling method was used while members of the research team were on shift. Subjects were informed of the study once they were triaged at the Emergency Department treatment area. Members were screened for pathological back pain by history and physical, and if negative were offered enrollment into the study. After informed consent and Health Insurance Portability and Accountability Act (HIPPA), demographics were collected as well as an initial Visual Analog Score (VAS) score, Numeric Rating Scale (NRS) score, and back pain functional scale (BPFS). Participants were randomly assigned to either the treatment or control group based on a random number generator. Subjects then received either BFA or the standard care, which was a pre-determined medicinal treatment. Participants were reassessed at 30-40 minutes post intervention for effectiveness of intervention for both pain and satisfaction. After initial pain control was achieved subjects completed a questionnaire on their perceived effectiveness of BFA as well as if they would repeat BFA in the future. If participants did not feel pain was adequately controlled in the either treatment arm they were provided rescue pain medications based on the preference of the treating provider. At discharge, participants were given further instructions including a follow-up telephone interview between 48-72 hours. In the telephone follow-up, participants were assessed on a Numerical Rating Scale (NRS), repeat functionality questionnaire, and if they used any other pain medications since discharge to help improve their pain (either pain medications given at discharge from the emergency department or their regularly prescribed pain medications).

Data Analysis: In this study, the independent variables were treatment for musculoskeletal pain in the emergency department (standard care, battlefield acupuncture) and time (before treatment, 30 to 40 minutes post-treatment and 48 to 72 hours post-treatment). The dependent variable is pain measured on a VAS or NRS at 48-72 hours post-treatment. The null hypothesis is that there is no statistically significant difference in pain related to treatment or time between treatment groups. With 26 subjects per group (52 total), the investigator was able to detect a 1.0 standard deviation (SD) difference measured by a 13mm change in the VAS or a 2 point change in the NRS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals to be enrolled the study will be:

  * Emergency Room patient
  * Able to provide informed consent (of sound mind)
  * acute defined as less than 3 months, or acute on chronic musculoskeletal pain
  * Individuals will be between 18-55 years of age and include Active Duty (AD) service members and beneficiaries
  * Pain at prescreening will be greater than or equal to 3 based on the Visual Analogue Scale (VAS).
  * Non-pathological acute back pain

Exclusion Criteria:

* The individuals eligible for the study will be in good health, as defined by the World Health Organization (WHO, 2006). "Health is a state of complete physical, mental, and social wellbeing and not merely the absence of disease or infirmity" (WHO, 2006). Specific exclusion criteria will include,

  * Participants presenting with open wound injuries
  * temperature >38.0 Celsius
  * suspected fractures
  * pain associated with diseases (flank/kidney pain)
  * concern for other than back pain (pyelonephritis, kidney stones, pathologic signs and symptoms)
  * bowel/bladder incontinence or retention
  * foot drop
  * known current/history of cancer
  * known bleeding disorders
  * active infection at the needled insertion site
  * If member is found to be pregnant at any time during screening process they will be removed from consideration before any treatment options are offered.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
time-response of BFA, and the association with pain level using the Visual Analog scale (0-10 mm) scoring as well as the Numeric Rating Scale (0-10) scoring | before treatment, 30-40 minutes post-treatment, and 48 to 72 hours post-treatment
  determine if there is any significant change in pain in the BFA treatment group at specific time points using the Visual Analog scale (0-10 mm) scoring as well as the Numeric Rating Scale (0-10) scoring
Evaluate the change of pain on Visual Analog scale (0-10mm) scoring with BFA administered in the emergency department for persons presenting with non-pathologic back pain. | baseline and at 30-40 minutes post treatment
  Using the Visual Analog scale which is a 10mm line, the patient will place a mark on the graph which will be measured to determine if there is any significant difference between the BFA treatment group pain at specific timepoints using the VAS. The lower the score determined on the scale corresponds to a lower pain level for the patient and a higher score corresponds to a higher pain level.
Evaluate the change of pain on Numeric Rating Scale (0-10) scoring with BFA administered in the emergency department for persons presenting with non-pathologic back pain. | baseline, 30-40 minutes, and 48-72 hours
  The Numeric Rating scale which is a scale that is verbally asked to determine the patients pain response on a scale from 0 to 10 determine if there is any significant difference between the BFA treatment group pain at specific timepoints using the NRS. The lower the score determined on the scale corresponds to a lower pain level for the patient and a higher score corresponds to a higher pain level.

SECONDARY OUTCOMES:
time-response | 30-40 minutes after treatment, and between 48-72 hours after discharge
  Time response will determine change in pain associated with the Numeric Rating scale (measured 0-10, 0 being least, 10 being most) from baseline, at 30-40 minutes after treatment, and between 48-72 hours after discharge.
Examine the functionality score changes at 3 time points using the Back Pain Functional Scale | baseline, at the time the patient is to be discharged from the Emergency Room (0-3 hrs post baseline assessment), and 48-72 hours after discharge
  Stratford et al developed the Back Pain Function Scale (BPFS) (scored 0-60 with higher scores showing no difficulty and lower scores showing patient is unable to perform activity) to evaluation functional ability in patients with back pain. The authors are from McMaster University Appalachian Physical Therapy (Georgia) and Virginia Commonwealth University.
Explore participant satisfaction of pain control in the BFA treatment group: 1 question | At discharge from the Emergency Room (0-3 hours post baseline assessment) and between 48-72 hours after discharge
  1 question regarding overall pain control satisfaction, and 2 specifically addressing those in the acupuncture group
The need for any additional pain medication outside of the treatment protocol | recorded at the 48-72 hours from discharge for the follow up interview
  Number of patients that required any additional pain medications either in the Emergency Room or at home to include over the counter or prescription

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bonjour, DSc, Principal Investigator — Program Director

REFERENCES:
- [Background] Buckenmaier CC 3rd, Rupprecht C, McKnight G, McMillan B, White RL, Gallagher RM, Polomano R. Pain following battlefield injury and evacuation: a survey of 110 casualties from the wars in Iraq and Afghanistan. Pain Med. 2009 Nov;10(8):1487-96. doi: 10.1111/j.1526-4637.2009.00731.x. Epub 2009 Oct 14. PMID 19843233
- [Background] Butler FK Jr, Kotwal RS, Buckenmaier CC 3rd, Edgar EP, O'Connor KC, Montgomery HR, Shackelford SA, Gandy JV, Wedmore I, Timby JW, Gross K, Bailey JA. A Triple-Option Analgesia Plan for Tactical Combat Casualty Care: TCCC Guidelines Change 13-04. J Spec Oper Med. 2014 Spring;14(1):13-25. doi: 10.55460/CBRW-A2G1. PMID 24604434
- [Background] Burns, S., et al. (2013). "Moving Acupuncture to the Frontline of Military Medical Care: A Feasibility Study." Medical Acupuncture 25(1): 49-54.
- [Background] Chang BH, Sommers E. Acupuncture and relaxation response for craving and anxiety reduction among military veterans in recovery from substance use disorder. Am J Addict. 2014 Mar-Apr;23(2):129-36. doi: 10.1111/j.1521-0391.2013.12079.x. Epub 2013 Aug 30. PMID 25187049
- [Background] Cohen SP, Griffith S, Larkin TM, Villena F, Larkin R. Presentation, diagnoses, mechanisms of injury, and treatment of soldiers injured in Operation Iraqi Freedom: an epidemiological study conducted at two military pain management centers. Anesth Analg. 2005 Oct;101(4):1098-1103. doi: 10.1213/01.ane.0000169332.45209.cf. PMID 16192528
- [Background] Corwell BN. The emergency department evaluation, management, and treatment of back pain. Emerg Med Clin North Am. 2010 Nov;28(4):811-39. doi: 10.1016/j.emc.2010.06.001. Epub 2010 Aug 4. PMID 20971393
- [Background] Delgado R, York A, Lee C, Crawford C, Buckenmaier C 3rd, Schoomaker E, Crawford P; Active Self-Care Therapies for Pain (PACT) Working Group. Assessing the quality, efficacy, and effectiveness of the current evidence base of active self-care complementary and integrative medicine therapies for the management of chronic pain: a rapid evidence assessment of the literature. Pain Med. 2014 Apr;15 Suppl 1:S9-20. doi: 10.1111/pme.12412. PMID 24734865
- [Background] Gawande A. Casualties of war--military care for the wounded from Iraq and Afghanistan. N Engl J Med. 2004 Dec 9;351(24):2471-5. doi: 10.1056/NEJMp048317. No abstract available. PMID 15590948
- [Background] Goertz CM, Niemtzow R, Burns SM, Fritts MJ, Crawford CC, Jonas WB. Auricular acupuncture in the treatment of acute pain syndromes: A pilot study. Mil Med. 2006 Oct;171(10):1010-4. doi: 10.7205/milmed.171.10.1010. PMID 17076456
- [Background] Gondusky JS, Reiter MP. Protecting military convoys in Iraq: an examination of battle injuries sustained by a mechanized battalion during Operation Iraqi Freedom II. Mil Med. 2005 Jun;170(6):546-9. doi: 10.7205/milmed.170.6.546. PMID 16001610
- [Background] Jones D, Shug S. Opioids in chronic pain of non-malignant origin: an interim consensus. N Z Med J. 1995 Nov 24;108(1012):492. No abstract available. PMID 8538981
- [Background] Kim KH, Lee BR, Ryu JH, Choi TY, Yang GY. The role of acupuncture in emergency department settings: a systematic review. Complement Ther Med. 2013 Feb;21(1):65-72. doi: 10.1016/j.ctim.2012.12.004. Epub 2012 Dec 29. PMID 23374207
- [Background] Lande RG. Sleep problems, posttraumatic stress, and mood disorders among active-duty service members. J Am Osteopath Assoc. 2014 Feb;114(2):83-9. doi: 10.7556/jaoa.2014.021. PMID 24481800
- [Background] Lazar SG. The mental health needs of military service members and veterans. Psychodyn Psychiatry. 2014 Sep;42(3):459-78. doi: 10.1521/pdps.2014.42.3.459. PMID 25211433
- [Background] Lew HL, Otis JD, Tun C, Kerns RD, Clark ME, Cifu DX. Prevalence of chronic pain, posttraumatic stress disorder, and persistent postconcussive symptoms in OIF/OEF veterans: polytrauma clinical triad. J Rehabil Res Dev. 2009;46(6):697-702. doi: 10.1682/jrrd.2009.01.0006. PMID 20104399
- [Background] Outcalt SD, Ang DC, Wu J, Sargent C, Yu Z, Bair MJ. Pain experience of Iraq and Afghanistan Veterans with comorbid chronic pain and posttraumatic stress. J Rehabil Res Dev. 2014;51(4):559-70. doi: 10.1682/JRRD.2013.06.0134. PMID 25144169
- [Background] Patel TH, Wenner KA, Price SA, Weber MA, Leveridge A, McAtee SJ. A U.S. Army Forward Surgical Team's experience in Operation Iraqi Freedom. J Trauma. 2004 Aug;57(2):201-7. doi: 10.1097/01.ta.0000133638.30269.38. PMID 15345962
- [Background] Pennick V, Liddle SD. Interventions for preventing and treating pelvic and back pain in pregnancy. Cochrane Database Syst Rev. 2013 Aug 1;(8):CD001139. doi: 10.1002/14651858.CD001139.pub3. PMID 23904227
- [Background] Pilkington K, Kirkwood G, Rampes H, Cummings M, Richardson J. Acupuncture for anxiety and anxiety disorders--a systematic literature review. Acupunct Med. 2007 Jun;25(1-2):1-10. doi: 10.1136/aim.25.1-2.1. PMID 17641561
- [Background] Schug SA, Zech D, Grond S, Jung H, Meuser T, Stobbe B. A long-term survey of morphine in cancer pain patients. J Pain Symptom Manage. 1992 Jul;7(5):259-66. doi: 10.1016/0885-3924(92)90059-q. PMID 1624812
- [Background] Seal KH, Shi Y, Cohen G, Cohen BE, Maguen S, Krebs EE, Neylan TC. Association of mental health disorders with prescription opioids and high-risk opioid use in US veterans of Iraq and Afghanistan. JAMA. 2012 Mar 7;307(9):940-7. doi: 10.1001/jama.2012.234. PMID 22396516
- [Background] Seal KH, Metzler TJ, Gima KS, Bertenthal D, Maguen S, Marmar CR. Trends and risk factors for mental health diagnoses among Iraq and Afghanistan veterans using Department of Veterans Affairs health care, 2002-2008. Am J Public Health. 2009 Sep;99(9):1651-8. doi: 10.2105/AJPH.2008.150284. Epub 2009 Jul 16. PMID 19608954
- [Background] Sharpe Potter J, Bebarta VS, Marino EN, Ramos RG, Turner BJ. Pain management and opioid risk mitigation in the military. Mil Med. 2014 May;179(5):553-8. doi: 10.7205/MILMED-D-13-00109. PMID 24806501
- [Background] Tan HJ, Lan Y, Wu FS, Zhang HD, Wu L, Wu X, Liang FR. [Auricular acupuncture for primary insomnia: a systematic review based on GRADE system]. Zhongguo Zhen Jiu. 2014 Jul;34(7):726-30. Chinese. PMID 25233674
- [Background] Vas J, Aranda-Regules JM, Modesto M, Aguilar I, Baron-Crespo M, Ramos-Monserrat M, Quevedo-Carrasco M, Rivas-Ruiz F. Auricular acupuncture for primary care treatment of low back pain and posterior pelvic pain in pregnancy: study protocol for a multicentre randomised placebo-controlled trial. Trials. 2014 Jul 16;15:288. doi: 10.1186/1745-6215-15-288. PMID 25027493
- [Background] Vas J, Aguilar I, Perea-Milla E, Mendez C. Effectiveness of acupuncture and related techniques in treating non-oncological pain in primary healthcare--an audit. Acupunct Med. 2007 Jun;25(1-2):41-6. doi: 10.1136/aim.25.1-2.41. PMID 17641567
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186